CLINICAL TRIAL: NCT04724044
Title: A Randomized Clinical Trial of Oral Clarithromycin in Community-acquired Pneumonia to Attenuate Inflammatory Responses and Improve Outcomes: the ACCESS Clinical Trial
Brief Title: Anti-inflammatory Action of Oral Clarithromycin in Community-acquired Pneumonia
Acronym: ACCESS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hellenic Institute for the Study of Sepsis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ACCESS; 2020-004452-15 (EudraCT Number)
Record Dates: First submitted 2021-01-20; First posted 2021-01-26 (Actual); Last update posted 2023-12-12 (Actual); Status verified 2023-12

CONDITIONS: Community-acquired Pneumonia; Sepsis; Inflammatory Response; Mortality; Biomarkers; SIRS
Keywords: Macrolides; Clarithromycin
MeSH Terms: conditions — Community-Acquired Pneumonia; Sepsis | interventions — Tablets; Clarithromycin

STUDY DESIGN:
Intervention Model Description: This is a prospective, 1:1 randomized, double-blind, placebo-controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator): These patients will be treated with 1 placebo tablet every 12 hours and intravenously with ceftriaxone or one β-lactam/β-lactamase combination as part of standard of care therapy indicated by the summary of product characteristics and according to bibliographic references. The total duration of treatment will be seven days.The dose regimen of ceftriaxone will be 2g once daily. The β-lactam/β-lactamase combination can be either amoxycilln/clavulanate or ampicillin/sulbactam or piperacillin/tazobactam. These may be administered three or four times daily and the dose is adjusted according to renal clearance. In case urinary antigen for Legionella spp is positive and/or Mycoplasma pneumoniae spp is isolated in sputum culture and/or in BioFire Respiratory FilmArray, patients will receive intravenously 400mg of moxifloxacin instead of ceftriaxone as part of standard of care therapy according to bibliographic references.
  Interventions: Drug: Tablets
- Clarithromycin (Active Comparator): These patients will be treated with 1 tablet of 500 mg of clarithromycin every 12 hours and intravenously with ceftriaxone or one β-lactam/β-lactamase combination as part of standard of care therapy indicated by the summary of product characteristics and according to bibliographic references. The total duration of treatment will be seven days.The dose regimen of ceftriaxone will be 2g once daily. The β-lactam/β-lactamase combination can be either amoxycilln/clavulanate or ampicillin/sulbactam or piperacillin/tazobactam. These may be administered three or four times daily and the dose is adjusted according to renal clearance. In case urinary antigen for Legionella spp is positive and/or Mycoplasma pneumoniae spp is isolated in sputum culture and/or in BioFire Respiratory FilmArray, patients will receive intravenously 400mg of moxifloxacin instead of ceftriaxone as part of standard of care therapy according to bibliographic references.
  Interventions: Drug: Clarithromycin 500mg

INTERVENTIONS:
Drug: Tablets — Oral tablets of similar appearance to active study drug
  Other Names: 2g of intravenous ceftriaxone or one β-lactam/β-lactamase combination(dose adjusted according to renal clearance) or 400mg of intravenous moxifloxacin
  Arms: Placebo
Drug: Clarithromycin 500mg — Oral tablets of 500mg of clarithromycin
  Other Names: 2g of intravenous ceftriaxone or one β-lactam/β-lactamase combination(dose adjusted according to renal clearance) or 400mg of intravenous moxifloxacin
  Arms: Clarithromycin

SUMMARY:
Traditional management of community-acquired pneumonia (CAP) relies on the prompt administration of antimicrobials that target the most common causative pathogens. Retrospective analysis of observational clinical studies in CAP showed that the addition of macrolides to standard antibiotic therapy conferred a significant survival benefit. The proposed benefit of macrolides is coming from their anti-inflammatory mode of action. An RCT that proves the attenuation of the high inflammatory burden of the host with CAP after addition of clarithromycin in the treatment regimen is missing. This RCT is aiming to prove that addition of oral clarithromycin to a β-lactam rapidly attenuates the high inflammatory burden of the host in CAP.

DETAILED DESCRIPTION:
Community-acquired pneumonia (CAP) is one of the most common bacterial infections and a leading cause of death globally since many patients deteriorate into sepsis and organ dysfunction. Traditional management relies on the prompt administration of antimicrobials that target the most common causative pathogens namely Streptococcus pneumoniae, Mycoplasma pneumoniae, Chlamydophila pneumoniae and Legionella pneumophila. Although there was some hesitancy in the former guidelines of the Infectious Diseases Society of America (IDSA) and of the American Thoracic Society (ATS) to suggest a clear-cut role of macrolides for the management of CAP, the new guidelines published by the ATS in 2019 clearly suggest for the management of all cases of CAP either treated as out-patients or as in-patients with a combination of β-lactam with macrolides.

The shift in the position of ATS expressed in the 2019 guidelines is coming from the growing body of evidence that the addition of a macrolide in the treatment regimen of CAP is accompanied by considerable survival benefit. This finding is mainly coming from the retrospective analysis of observational clinical studies in CAP. Results were also supported by the meta-analysis of these studies . Superiority coming from the macrolide use is mainly shown in cases of severe CAP i.e. situations with pneumonia severity index (PSI) greater than 2 that are most commonly caused by S.pneumoniae. The proposed benefit of macrolides is coming from their anti-inflammatory mode of action. This statement generates two main questions: a) what an anti-inflammatory mode of action consists of in the clinical setting; and b) is this a common property for all macrolides? Although it is easy to suggest that an antimicrobial modulates immune responses in vitro, it is extremely difficult to prove this in vivo. The main hurdle is coming from the fact that it is difficult to decipher to what extent clinical benefit is coming from the antimicrobial effect per se and to what extent this is due to modulation of the immune responses. In other terms, an anti-inflammatory effect is better shown in infections caused by pathogens that do not belong to the antimicrobial spectrum of macrolides. Our group has conducted two large scale randomized clinical trials (RCTs) where clarithromycin was co-administered intravenously along with β-lactams in either patients with ventilator-associated pneumonia (VAP) by multidrug-resistant Gram-negative pathogens or patients with severe Gram-negative infections like acute pyelonephritis, intraabdominal infections and primary Gram-negative bacteremia. The total number of patients enrolled in both studies was 800 and isolated pathogens did not belong to the antimicrobial spectrum of macrolides. Addition of clarithromycin provided overall survival benefit after 90-days in patients with VAP (57% survival versus 40% of placebo-treated comparators). Mortality by septic shock after 28-days was also considerably decreased in patients with severe Gram-negative infections (53.1% versus 73.1% of the comparators).

Although these findings point towards an anti-inflammatory mode of action of clarithromycin, they do not necessarily imply that a survival benefit similar to Gram-negative infections will apply in CAP. There is only one RCT to test the anti-inflammatory effect of clarithromycin in patients with CAP. This RCT was designed for non-inferiority and randomized patients were allocated into single β-lactam treatment or the combination with oral clarithromycin. The primary endpoint was clinical instability after seven days. Contrary to what investigators were expecting this was shown in 41.2% of non-macrolide treated patients and 33.6% of macrolide-treated patients (p: 0.070). It may be argued that if the study was powered for superiority, the study primary endpoint would have shown benefit from the addition of clarithromycin.

In recent publication coming from the research network of the Hellenic Sepsis Study Group (HSSG) 130 patients with CAP were treated with a combination of β-lactam and clarithromycin. They were compared with another 130 patients treated with a combination of β-lactam and azithromycin, with 130 patients treated with respiratory fluoroquinolone monotherapy and with 130 treated with β-lactam monotherapy. The study has a case-matching design and selection of cases of the three comparator groups were based on the group of patients treated with clarithromycin. Matching selection criteria were severity as assessed by the severity score of SOFA (sequential organ failure assessment), APACHE II (acute physiology and chronic health evaluation), PSI and CCI (Charlson's comorbidity index) and type of β-lactam. The 28-day mortality of the four groups was 20.8%, 33.8%, 32.3% and 36.2% respectively, showing a profound survival benefit with the intake of clarithromycin.

Based on the above analysis, it seems likely that an RCT that proves the attenuation of the high inflammatory burden of the host with CAP after addition of clarithromycin in the treatment regimen is missing. The need for this RCT is outscored in the recent guidelines of ATS . Such a type of RCT should take into consideration the SOFA score of the patients, the presence of the systemic inflammatory response syndrome (SIRS), the existence of elevated procalcitonin (PCT) in serum and the outcome of patients infected by macrolide-resistant S.pneumoniae. SOFA score is nowadays proposed as the sine qua non for severity. PCT more than 0.25 ng/ml is widely accepted as an index of systemic inflammation in the event of CAP to such an extent that decrease more than 80% or to levels lower than 0.25 ng/ml can be used as an index of therapy withdrawal. In such an RCT rapid resolution of the high inflammatory burden of the host should be highlighted in the achievement of the early treatment response of CAP after 72 hours that is recently appointed by the Food and Drug Administration and the European Medicines Agency as the primary endpoint goal of CAP.

This is an RCT that is aiming to prove that addition of oral clarithromycin to a β-lactam rapidly attenuates the high inflammatory burden of the host in CAP.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥18 years)
* Male of female gender
* In case of non-menopausal women, unwillingness to become pregnant during the study period. Women of child-bearing potential will be screened by a urine pregnancy test before inclusion in the study.
* Written informed consent provided by the patients or by a first-degree relative in case of patients unable to consent
* Presence of at least two signs of SIRS (see below for definition)
* SOFA score ≥2 (see Appendix I)
* PCT ≥0.25 ng/ml
* Presence of at least two of the following signs: i) cough; ii) purulent sputum expectoration; iii) dyspnea; and/or iv) pleuritic chest pain
* Presence of CAP (see below for definition)

SIRS is defined by the presence of at least two of the following criteria:

* Core temperature >38 Celsius degrees or <36 Celsius degrees
* Heart rate >90 beats/minute
* Breath rate >20 breaths/minute or pco2<32 mmHg
* Total white blood cell count >12,000/mm3 or <4,000/mm3 or >15% bands

CAP is defined as the presence of auscultatory findings compatible with CAP and new consolidation in chest X-ray in a patient without any history of contact with the hospital environment or with health-care facilities the last 90 days.

Exclusion Criteria:

* Age below 18 years
* Denial of written informed consent
* Presence of infection by SARS-CoV-2 (COVID-19)
* Intake of any macrolide for the current episode of CAP under study
* Oral or intravenous intake of corticosteroids defined as any more than 0.4mg/kg daily intake of equivalent prednisone for the last 15 days
* Neutropenia defined as an absolute neutrophil count below 1,000/mm3
* Known infection by the human immunodeficiency virus
* Any chronic anti-cytokine treatment (e.g. antibodies against TNF for rheumatoid arthritis)
* Hospitalization for more than 2 days the last 90 days
* QTc interval at rest ECG ≥500 msec or history of known congenital long QT syndrome
* Concomitant administration with HMG-CoA reductase inhibitors (statins) that are extensively metabolized by CYP3A4, (lovastatin or simvastatin), and presence of any contraindications for the study drug
* Pregnancy or lactation. Women of child-bearing potential will be screened by a urine pregnancy test before inclusion in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 278 (Actual)
Dates: Start 2021-01-25 (Actual); Primary Completion 2023-04-11 (Actual); Study Completion 2023-04-11 (Actual)

PRIMARY OUTCOMES:
Change of baseline respiratory symptoms score | 4 days
  At least 50 percent (%) decrease of the sum of scoring (0-12) for the symptoms of cough (0-3), dyspnea (0-3), purulent sputum expectoration (0-3) and pleuritic chest pain (0-3) between baseline and Study Day 4
Change of baseline total sequential organ failure assessment (SOFA) score and/or change of baseline serum PCT | 4 days
  At least 30 percent (%) decrease between baseline sequential organ failure assessment (SOFA) score and measured sequential organ failure assessment (SOFA) score at Study Day 4 and/or at least 80 percent (%) decrease of serum PCT from baseline PCT at Study Day 4 and/or serum PCT below 0.25 ng/ml at Study Day 4

SECONDARY OUTCOMES:
Change of baseline respiratory symptoms score in the subgroup of patients infected or colonized by clarithromycin-susceptible S.pneumoniae | 4 days
  Comparison of the number of patients reaching at least 50 percent (%) decrease of the sum of scoring (0-12) for the symptoms of cough (0-3), dyspnea (0-3), purulent sputum expectoration (0-3) and pleuritic chest pain (0-3) between baseline and Study Day 4, among clarithromycin and placebo-treated patients, infected or colonized by clarithromycin-susceptible S.pneumoniae
Change of baseline respiratory symptoms score in the subgroup of patients infected or colonized by clarithromycin-resistant S.pneumoniae | 4 days
  Comparison of the number of patients reaching at least 50 percent (%) decrease of the sum of scoring (0-12) for the symptoms of cough (0-3), dyspnea (0-3), purulent sputum expectoration (0-3) and pleuritic chest pain (0-3) between baseline and Study Day 4, among clarithromycin and placebo-treated patients, infected or colonized by clarithromycin-susceptible S.pneumoniae
Change of baseline total sequential organ failure assessment (SOFA) score and/or change of baseline serum PCT in the subgroup of patients infected or colonized by clarithromycin-susceptible S.pneumoniae | 4 days
  Comparison of the number of patients reaching at least 30 percent (%) decrease between baseline sequential organ failure assessment (SOFA) score and measured sequential organ failure assessment (SOFA) score at Study Day 4 and/or at least 80 percent (%) decrease of serum PCT from baseline at Study Day 4 and/or serum PCT below 0.25 ng/ml at Study Day 4, among clarithromycin and placebo-treated patients infected or colonized by clarithromycin-susceptible S.pneumoniae
Change of baseline total sequential organ failure assessment (SOFA) score and/or change of baseline serum PCT in the subgroup of patients infected or colonized by clarithromycin-resistant S.pneumoniae | 4 days
  Comparison of the number of patients reaching at least 30 percent (%) decrease between baseline sequential organ failure assessment (SOFA) score and measured sequential organ failure assessment (SOFA) score at Study Day 4 and/or at least 80 percent (%) decrease of serum PCT from baseline at Study Day 4 and/or serum PCT below 0.25 ng/ml at Study Day 4, among clarithromycin and placebo-treated patients infected or colonized by clarithromycin-resistant S.pneumoniae
Mortality rate at 28 days | 28 days
  Differences in 28-day all-cause mortality rate between clarithromycin and placebo-treated arms
Mortality rate at 90 days | 90 days
  Differences in 90-day all-cause mortality rate between clarithromycin and placebo-treated arms
Clinical success at the end of treatment Visit (day 8) | 8 days
  Difference in clinical success rate at day 8, as defined by at least 50 percent (%) decrease of the baseline sum of scoring (0-12) for the symptoms of cough (0-3), dyspnea (0-3), purulent sputum expectoration (0-3) and pleuritic chest pain (0-3)
Hospital discharge until day 90 | 90 days
  Comparison of length of hospital stay (days) until day 90 between clarithromycin and placebo-treated arms
Hospital readmission until day 90 | 90 days
  Comparison of hospital readmission rate until day 90 between clarithromycin and placebo-treated arms
Change of baseline total sequential organ failure assessment (SOFA) score at the end of treatment Visit (day 8) | 8 days
  Comparison of number of patients reaching more than 50 percent (%) decrease between baseline sequential organ failure assessment (SOFA) score and measured sequential organ failure assessment (SOFA) score at Study Day 8 between clarithromycin and placebo-treated arms
Development of new organ dysfunctions until day 90 | 90 days
  Comparison of the rate of development of new organ dysfunctions between clarithromycin and placebo-treated arms
Change of function of monocytes, Th1, Th2 and T17 cells at Study Visit 4 | 4 days
  Comparison of cytokine production by stimulation of monocytes, Th1,Th2 and T17 cells between clarithromycin and placebo-treated arms
Change of gene expression of anti-inflammatory genes at Study Visit 4 | 4 days
  Comparison of the expressions of four genes (FGL-2, IL7R, HLA-DPA1, CPVL), that are down-regulated upon development of severe infections, between clarithromycin and placebo-treated arms
Anti-inflammatory PCT change at study Visit 6 | 6 days
  Comparison of number of patients reaching at least 80 percent (%) decrease of serum PCT from baseline on day 6 or any value of PCT below 0.25 ng/ml on day 6 between clarithromycin and placebo-treated arms
Anti-inflammatory PCT change at the end of treatment Visit (day 8) | 8 days
  Comparison of number of patients reaching at least 80 percent (%) decrease of serum PCT from baseline on day 8 or any value of PCT below 0.25 ng/ml on day 8 between clarithromycin and placebo-treated arms
Change of the IL-10/TNFα ratio at study Visit 6 | 6 days
  Comparison of the change of the IL-10/TNFα ratio between baseline and day 6 among clarithromycin and placebo-treated arms
Change of the IL-10/TNFα ratio at the end of treatment Visit (day 8) | 8 days
  Comparison of the of the change of the IL-10/TNFα ratio between baseline and day 8 among clarithromycin and placebo-treated arms
New sepsis episode until day 90 | 90 days
  Comparison of the rate of development of new sepsis episode between clarithromycin and placebo-treated arms
Change of expression of the MVK gene at study Visit 4 | 4 days
  Comparison of the expression of the MVK gene, that affects the cholesterol homeostasis pathway, between clarithromycin and placebo-treated arms
Change of expression of the SC5D gene at study Visit 4 | 4 days
  Comparison of the expression of the SC5D gene, that affects the cholesterol homeostasis pathway, between clarithromycin and placebo-treated arms
Change of expression of the MVD gene at study Visit 4 | 4 days
  Comparison of the expression of the MVD gene, that affects the cholesterol homeostasis pathway, between clarithromycin and placebo-treated arms
Change of expression of the STARD4 gene at study Visit 4 | 4 days
  Comparison of the expression of the STARD4 gene, that affects the cholesterol homeostasis pathway, between clarithromycin and placebo-treated arms
Change of expression of the SQLE gene at study Visit 4 | 4 days
  Comparison of the expression of the SQLE gene, that affects the cholesterol homeostasis pathway, between clarithromycin and placebo-treated arms

CONTACTS AND LOCATIONS:
Overall Officials: Evangelos J Giamarellos-Bourboulis, MD, PhD, Study Chair — Hellenic Sepsis Study Group
Locations (18):
- Greece (18):
  - 4th Department of Internal Medicine, Attikon University Hospital, Athens
  - 1st Department of Internal Medicine, Amalia Fleming General Hospital, Athens
  - 1st Department of Internal Medicine, Gennimatas General Hospital, Athens
  - 1st Department of Internal Medicine, Konstantopouleio-Patission General Hospital, Athens
  - 1st Department of Internal Medicine, THRIASIO Eleusis General Hospital, Athens
  - 1st Department of Internal Medicine,Korgialeneio-Benakeio General Hospital, Athens
  - 2nd Department of Internal Medicine, Attikon University Hospital, Athens
  - 2nd Department of Internal Medicine, Thriasio General Hospital, Athens
  - 3rd Department of Internal Medicine, KORGIALENEION-BENAKEION Athens General Hospital, Athens
  - 3rd Department of Internal Medicine, Sotiria General Hospital, Athens
  - 5th Department of Internal Medicine, Evangelismos General Hospital, Athens
  - Department of Chest Medicine, EVANGELISMOS Athens General Hospital, Athens
  - Department of Pulmonary Medicine, General Hospital of Kerkyra, Corfu
  - 1st Department of Internal Medicine, Ioannina University General Hospital, Ioannina
  - Department of Internal Medicine, Larissa University General Hospital, Larissa
  - Department of Internal Medicine, Patras University General Hospital, Pátrai
  - 2nd Department of Internal Medicine, Tzaneion General Hospital, Piraeus
  - Department of Emergency Medicine, Tzanneion General Hospital, Piraeus

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Giamarellos-Bourboulis EJ, Siampanos A, Bolanou A, Doulou S, Kakavoulis N, Tsiakos K, Katopodis S, Schinas G, Skorda L, Alexiou Z, Armenis K, Katsaounou P, Chrysos G, Masgala A, Poulakou G, Antonakos N, Safarika A, Kyprianou M, Dakou K, Gerakari S, Papanikolaou IC, Milionis H, Marangos M, Dalekos GN, Tzavara V, Akinosoglou K, Hatziaggelaki E, Sympardi S, Kontopoulou T, Mouktaroudi M, Papadopoulos A, Niederman MS. Clarithromycin for early anti-inflammatory responses in community-acquired pneumonia in Greece (ACCESS): a randomised, double-blind, placebo-controlled trial. Lancet Respir Med. 2024 Apr;12(4):294-304. doi: 10.1016/S2213-2600(23)00412-5. Epub 2024 Jan 3. PMID 38184008